CLINICAL TRIAL: NCT05578768
Title: Prediction of IBD Disease Activity in Individual Patients Based on PROMs and Clinical Data
Acronym: PrePro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Alrijne Hospital (Other); Maasstad Hospital (Other)
Responsible Party: Principal Investigator, Andrea E. van der Meulen - de Jong, MD, PhD, Principal Investigator, Leiden University Medical Center
Other Study IDs: nWMODIV2_2022020
Record Dates: First submitted 2022-08-17; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: IBD; Inflammatory Bone Disease
MeSH Terms: conditions — Osteitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training phase: The study procedures for both cohorts are the same.
  Interventions: Other: No intervention
- validation phase: The study procedures for both cohorts are the same.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Patients will receive standard of care.

SUMMARY:
The proposed study will use a PROM (Patient report Outcome Measurement)-tool in combination with clinical and biochemical data to train and validate a Relapse Prediction Model for individual patients.

DETAILED DESCRIPTION:
The primary objective is to train and validate a relapse prediction model for individual patients available for daily (remote) care management. Besides that, risk-based care pathways for different prediction outcomes will be evaluated, prediction scores will be correlated to medication type, CRP/Calprotectin and/or endoscopy, and with known IBD clinical risk profiles. Moreover dietary intake will be correlated with the IBD risk profiles.

Study design: Multicentre, retrospective analysis of two prospective cohorts. Study population: Adult IBD patients. Main study parameters/endpoints: The endpoint will be a prediction regarding step-up or step-down in the care pathways. In other words, the percentage of patients in each individual care pathway with agreement between risk score of the individual patient and actual flares during a follow-up time of 24 months. Furthermore insight will be gained in dietary patterns amongst patients with different IBD risk profiles.

No benefits or risks are associated with participating in this study, because only standard of care is given.

ELIGIBILITY:
Inclusion Criteria:

* Adult IBD patients
* Subjects willing and able to sign informed consent
* Own and are able to use a smart phone (Android or iOS)

Exclusion Criteria:

* Unwilling or unable to adhere to the protocol
* Unwilling or unable to adhere to the informed consent
* Age <18y

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In clinical practice, consecutive IBD patients in the LUMC, AH, and MH are registered on the platform and will be asked to participate in the current project. At least 200 UC patients and at least 200 CD patients will be included. Following inclusion, each patient will spend at least 12, but preferably 24 months on the platform.
  Patients are already using the PROM-tool to allow remote monitoring; this has been implemented since 2021.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Develop a relapse prediction model for individual patients (agreement between risk score of the individual patient and actual flares) based on both clinical parameters and biochemical parameters in the individual care pathways. | After 2 years
  This model will be based on both clinical parameters and biochemical parameters in the individual care pathways.
Validate the above mentioned prediction model and make it available for daily (remote) care management. | After 2 years
  Based on the information form the validation cohort. The model will be validated retrospectively.

SECONDARY OUTCOMES:
evaluate risk-based care pathways for different prediction outcomes in clinical practice e.g. high intensity monitoring care pathway for patients with a high prediction score. | After 2 years
  Evaluate whether predefined risk-based care pathways are in line with prediction outcomes of the relapse prediction model.
Correlate the prediction scores of the different care pathways to medication type. | After 2 years
  See if there is a statistical correlation between medication type and prediction score
Correlate prediction scores of the different pathways with biomarkers CRP/Calprotectin and/or endoscopy | After 2 years
  See if there is a statistical correlation between prediction score and biomarkers CRP/Calprotectin and/or endoscopy
Correlate prediction scores from the algorithm with known IBD clinical risk factors | After 2 years
  See if there is a statistical correlation between prediction scores from the model to known clinical risk factors like e.g. operation history, presence of EIM.
Correlate dietary intake with the assigned IBD clinical risk profiles | After 2 years
  See if there is a statistical correlation between dietary intake and assigned IBD clinical risk profile.

CONTACTS AND LOCATIONS:
Overall Officials: A.E. van der Meulen - de Jong, MD, PhD, Principal Investigator — Leiden University Medical Centre
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands